CLINICAL TRIAL: NCT00421434
Title: Randomized Study of Nitazoxanide-Peginterferon, Nitazoxanide-Peginterferon-Ribavirin and Peginterferon-Ribavirin in the Treatment of Chronic Hepatitis C
Brief Title: Study of Nitazoxanide, Peginterferon, and Ribavirin Combination Therapies in the Treatment of Chronic Hepatitis C
Acronym: STEALTHC-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Romark Laboratories, L.C., Romark Laboratories, L.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM01-3036
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — nitazoxanide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nitazoxanide-Peginterferon (Experimental): One oral nitazoxanide 500 mg tablet with food twice daily for 12 weeks followed by 36 weeks of one oral nitazoxanide 500 mg tablet plus weekly injections of 180 µg peginterferon alfa-2a.
  Interventions: Drug: Nitazoxanide; Biological: Peginterferon alfa-2a
- Nitazoxanide-Peginterferon-Ribavirin (Experimental): One oral nitazoxanide 500 mg tablet with food twice daily for 12 weeks followed by 36 weeks of one oral nitazoxanide 500 mg tablet plus weekly injections of 180 µg peginterferon alfa-2a plus oral ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight ≥75 kg) daily in two divided doses.
  Interventions: Drug: Nitazoxanide; Biological: Peginterferon alfa-2a; Drug: Ribavirin
- Peginterferon-Ribavirin (Active Comparator): Weekly injections of 180 µg peginterferon alfa-2a plus oral ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight ≥75 kg) daily in two divided doses for 48 weeks.
  Interventions: Biological: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Nitazoxanide — One oral nitazoxanide 500 mg tablet with food twice daily for 48 weeks.
  Other Names: Alinia
  Arms: Nitazoxanide-Peginterferon; Nitazoxanide-Peginterferon-Ribavirin
Biological: Peginterferon alfa-2a — Weekly injections of 180µg peginterferon alfa-2a for 36 weeks.
  Other Names: PEGASYS
  Arms: Nitazoxanide-Peginterferon; Nitazoxanide-Peginterferon-Ribavirin
Biological: Peginterferon alfa-2a — Weekly injections of 180 µg peginterferon alfa-2a for 48 weeks.
  Other Names: PEGASYS
  Arms: Peginterferon-Ribavirin
Drug: Ribavirin — Oral ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight ≥75 kg) daily in two divided doses for 36 weeks.
  Other Names: COPEGUS
  Arms: Nitazoxanide-Peginterferon-Ribavirin
Drug: Ribavirin — Oral ribavirin 1000 mg (body weight <75 kg) or 1200 mg (body weight ≥75 kg) daily in two divided doses for 48 weeks.
  Other Names: COPEGUS
  Arms: Peginterferon-Ribavirin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nitazoxanide-peginterferon and nitazoxanide-peginterferon-ribavirin combination regimens compared to the standard of care (peginterferon-ribavirin) in treating chronic hepatitis C genotype 4. The study will also evaluate the effect of the studied treatment regimens on end of treatment virologic response, ALT normalization and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Chronic hepatitis C infection (at least 6 months) evidenced by a positive enzyme immunoassay for anti-HCV-antibodies and a positive quantitative RT-PCR amplification of HCV RNA.
* Chronic inflammation on liver biopsy compatible with a diagnosis of chronic viral hepatitis.
* HCV genotype 4.

Exclusion Criteria:

* Patients who have previously failed to respond to ≥12 weeks of peginterferon-ribavirin combination therapy.
* Females who are either pregnant, breast-feeding or not using birth control and are sexually active.
* Males whose female partners are pregnant.
* Patients with other causes of liver disease (i.e., autoimmune hepatitis, decompensated liver disease).
* Patients co-infected with hepatitis A virus, hepatitis B virus or hepatitis D virus.
* Patients with a history of alcoholism or with an alcohol consumption of >40 grams per day.
* Patients with hemoglobinopathies (i.e., thalassemia major, sickle-cell anemia).
* Patients with any concomitant condition that, in the opinion of the investigator, would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed.
* History of hypersensitivity or intolerance to any of the excipients comprising the nitazoxanide tablets, peginterferon alfa-2a injectionable solution or ribavirin tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response | 24 weeks after the end of treatment

SECONDARY OUTCOMES:
End of treatment virologic response | At the end of treatment
Early virologic response | After 12 weeks of combination therapy
Rapid virologic response | After 4 weeks of combination therapy
ALT normalization | 24 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yehia El-Gohary, MD, Principal Investigator — Department of Tropical Medicine & Infectious Diseases, Alexandria University; Asem Elfert, MD, Principal Investigator — Department of Tropical Medicine & Infectious Diseases, Tanta University School of Medicine
Locations (2):
- Egypt (2):
  - Department of Tropical Medicine & Infectious Diseases, Alexandria University, Alexandria
  - Department of Tropical Medicine & Infectious Diseases, Tanta University School of Medicine, Tanta